CLINICAL TRIAL: NCT04779112
Title: Detecting Acetabulum Movement After Total Hip Arthroplasty From Serial Plain Radiographs
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: N201912060
Record Dates: First submitted 2021-02-22; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Orthopedics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study mainly measures the orientation of acetabulum cup post total hip arthroplasty. Using "Liaw's Version", a new and accurate standardization method, investigators are trying to analyze acetabulum cup anterversion change postoperatively.

DETAILED DESCRIPTION:
Patients undergoing total hip arthroplasty have generally good prognosis. However, clinically there was still a minority of patients who suffered from persistent postoperative pain. Dislocations of hip leading to revision surgeries were as well observed in some patients.

This study mainly measures the orientation of acetabulum cup post total hip arthroplasty. Using "Liaw's Version", a new and accurate standardization method, investigators are trying to analyze acetabulum cup anterversion change postoperatively.

As previously known, the anteversion of acetabulum cup determines the range of motion, stability, and the function after total hip arthroplasty. Cup malalignment increase impingement, dislocation, cup migration, and polyethylene wear. Finding a pattern may help the early diagnosis of acetabular loosening.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergone total hip arthroplasty
* Patients undergone total hip arthroplasty with more than two postoperative X-ray plain films

Exclusion Criteria:

* Patients with postoperative periprosthetic fracture(s)
* Patients with postoperative infection
* Patients undergone revision total hip arthroplasty

Ages: 40 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients of hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Analyze acetabulum cup anterversion change postoperatively | 1 week
  Using "Liaw's Version", a new and accurate standardization method developed, investigators are trying to analyze acetabulum cup anterversion change postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Kun Liaw, Study Chair — Taipei Medical University